CLINICAL TRIAL: NCT04568785
Title: Effectiveness of a Brief Intervention for Acceptance of Influenza Vaccine in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Principal Investigator, Raquel Muñoz Miralles, Primary Health Care Nurse, Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P17/224
Record Dates: First submitted 2020-09-14; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Influenza Vaccination; Health Education
Keywords: directive counseling; health education; influenza vaccines; primary health care; vaccination coverage
MeSH Terms: conditions — Influenza, Human; Health Education | interventions — Crisis Intervention; Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intervention group (Experimental): Intervention consisted of a standardized Brief Intervention, which varied depending on the reason the patient had given for refusing the vaccination.
  Interventions: Behavioral: Brief Intervention for Influenza vaccine
- Control group (Active Comparator): the control group intervention was the normal advice that professionals used to give their patients
  Interventions: Behavioral: Normal advice

INTERVENTIONS:
Behavioral: Brief Intervention for Influenza vaccine — Previous to the intervention, patients were asked about the reasons to reject the influenza vaccine. Brief Intervention was performed by the healthcare professional during the consultation. It was given verbally, with written support.
  Arms: Brief Intervention group
Behavioral: Normal advice — In the CG the influenza vaccine advice was the normal advice that professionals used to give their patients and was not asked for the reasons for the rejection of the vaccine to prevent them from influencing the advice.
  Arms: Control group

SUMMARY:
Influenza virus has high morbidity rates during annual epidemics, with certain high-risk groups being particularly susceptible to complications and mortality. Vaccination is the main prevention measure, alongside with hygiene measures. Nevertheless, vaccine coverage remains low.

Some studies suggest that short, standardized interventions can improve coverage of several vaccines.

Hypothesis: Brief Intervention is an effective tool in improving vaccination coverage in people who have initially rejected it.

Objective: To determine the effectiveness of a Brief Intervention in increasing influenza vaccination (IIV) coverage compared with the usual advice in people who refuse it.

Method: cluster randomized clinical trial. The study population was individuals with high risk factors who initially refused the influenza vaccine. Professionals participants (doctors and nurses) were assigned randomly to the intervention group (brief intervention) and the control group (usual advice).

DETAILED DESCRIPTION:
General objective: To determine the effectiveness of the use of BI for IIV compared to the usual advice, in people who refuse to be vaccinated.

Specific objectives:

1. To examine the effectiveness of Brief Intervention compared to the usual advice in different risk groups (> 60 healthy, > 60 years old with a Risk Factor [RF], <60 years old with RF).
2. Quantify influenza vaccine coverage in people with the most frequent RF.
3. Record the patients' reasons for refusing to be vaccinated.

METHOD A cluster randomized controlled clinical trial. The reference population consisted of patients assigned to and treated by urban and rural health centres in the centre of Catalonia, an area with a population of approximately 405,000. 135,648 were the risk factor population that could be vaccinated against influenza virus.

The study population consisted of individuals with high risk factors who were treated in healthcare centres during the 2017 influenza campaign.

The study protocol was approved by the Research Ethics Committee (CEI) of the Institut Universitari d'Investigació en Atenció Primària (IDIAP Jordi Gol).

The participants (doctors and nurses) decided voluntarily whether or not to participate and they were randomly assigned to either the Intervention Group (IG) or the Control Group (CG).

The recruitment of patients suitable to participate in the study was carried out during the IIV campaign, as part of the health centre's routine activities. Patients with inclusion criteria who came to see a doctor or nurse were invited to participate in the study. Those who accepted participating signed an informed consent.

The intervention consisted of a standardized Brief Intervention for the Influenza Vaccination.

Data was collected anonymously and confidentially via the electronic health record of Catalonia [eCAP in Catalan]. The variables analysed for the two groups were: IIV at the end of the 2017 vaccination campaign (yes/no), age, IIV risk factors and reasons for non-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Individuals in high-risk groups for influenza (paediatric and adult)
* Not intending to be vaccinated against the influenza virus during the current season.
* Informed consent to participate. In case of paediatric patients, parents signed the consent and made decisions about vaccination.

Exclusion Criteria:

* Language barrier
* Mental or physical conditions which make it difficult for the patient or their relatives to make decisions.
* Having previously participated in the pilot study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 524 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
Influenza vaccination status at the end of the Influenza vaccination campaign 2017. | up to 3 months
  % of reluctant patients vaccinated against Influenza at the end of the campaign 2017. Measurement tool: Influenza vaccine registered in patient's medical history
Influenza vaccination status of the participants who received the Brief Intervention or the normal advice. | up to 3 months
  % of reluctant patients vaccinated against Influenza in the Intervention group or in the Control group. Measurement tool: Influenza vaccine registered in patient's medical history

SECONDARY OUTCOMES:
Reasons for rejecting Influenza Vaccination | one day
  % of the different reasons for rejecting Influenza Vaccination. Measurement tool: specific questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- CAP Plaça Catalunya- Manresa 2, Manresa, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bish A, Yardley L, Nicoll A, Michie S. Factors associated with uptake of vaccination against pandemic influenza: a systematic review. Vaccine. 2011 Sep 2;29(38):6472-84. doi: 10.1016/j.vaccine.2011.06.107. Epub 2011 Jul 12. PMID 21756960
- [Background] Giese C, Mereckiene J, Danis K, O'Donnell J, O'Flanagan D, Cotter S. Low vaccination coverage for seasonal influenza and pneumococcal disease among adults at-risk and health care workers in Ireland, 2013: The key role of GPs in recommending vaccination. Vaccine. 2016 Jul 12;34(32):3657-62. doi: 10.1016/j.vaccine.2016.05.028. Epub 2016 Jun 7. PMID 27255466
- [Background] Picazo J, González Romo F, Salleras Sanmartí J, Bayas Rodríguez J, Álvarez Pasquín M. Encuesta sobre la vacunación de adultos en España. Gripe y neumococo. Vacunas. 2012; 13(3): 100-111. doi.10.1016/S1576-9887(12)70048-1
- [Background] Stockwell MS, Kharbanda EO, Martinez RA, Vargas CY, Vawdrey DK, Camargo S. Effect of a text messaging intervention on influenza vaccination in an urban, low-income pediatric and adolescent population: a randomized controlled trial. JAMA. 2012 Apr 25;307(16):1702-8. doi: 10.1001/jama.2012.502. PMID 22535855
- [Background] European Centre for Disease Prevention and Control. Catalogue of interventions addressing vaccine hesitancy. Stockholm: ECDC; 2017. doi: 10.2900/654210
- [Background] Whitlock EP, Orleans CT, Pender N, Allan J. Evaluating primary care behavioral counseling interventions: an evidence-based approach. Am J Prev Med. 2002 May;22(4):267-84. doi: 10.1016/s0749-3797(02)00415-4. PMID 11988383
- [Background] Wong VW, Fong DY, Tarrant M. Brief education to increase uptake of influenza vaccine among pregnant women: a study protocol for a randomized controlled trial. BMC Pregnancy Childbirth. 2014 Jan 14;14:19. doi: 10.1186/1471-2393-14-19. PMID 24423245
- [Background] Wong VWY, Fong DYT, Lok KYW, Wong JYH, Sing C, Choi AY, Yuen CYS, Tarrant M. Brief education to promote maternal influenza vaccine uptake: A randomized controlled trial. Vaccine. 2016 Oct 17;34(44):5243-5250. doi: 10.1016/j.vaccine.2016.09.019. Epub 2016 Sep 22. PMID 27667330
- [Background] Ferguson PE, Jordens CF, Gilroy NM. Patient and family education in HSCT: improving awareness of respiratory virus infection and influenza vaccination. A descriptive study and brief intervention. Bone Marrow Transplant. 2010 Apr;45(4):656-61. doi: 10.1038/bmt.2009.209. Epub 2009 Aug 17. PMID 19684629
- [Background] Chan SS, Leung DY, Leung AY, Lam C, Hung I, Chu D, Chan CK, Johnston J, Liu SH, Liang R, Lam TH, Yuen KY. A nurse-delivered brief health education intervention to improve pneumococcal vaccination rate among older patients with chronic diseases: a cluster randomized controlled trial. Int J Nurs Stud. 2015 Jan;52(1):317-24. doi: 10.1016/j.ijnurstu.2014.06.008. Epub 2014 Jun 19. PMID 25012957
- [Background] Bonafide KE, Vanable PA. Male human papillomavirus vaccine acceptance is enhanced by a brief intervention that emphasizes both male-specific vaccine benefits and altruistic motives. Sex Transm Dis. 2015 Feb;42(2):76-80. doi: 10.1097/OLQ.0000000000000226. PMID 25585065
- [Background] Muñoz-Miralles R, Bonvehí Nadeu S, Sant Masoliver C, Martín Gallego A, Llamazares Robles MO, Mendioroz Peña J. Efectividad del consejo breve en la vacunación contra la gripe. Estudio piloto en atención primaria. Vacunas. 2019; 20(1): 18-24. doi.10.1016/j.vacun.2019.01.001
- [Background] Nyhan B, Reifler J. Does correcting myths about the flu vaccine work? An experimental evaluation of the effects of corrective information. Vaccine. 2015 Jan 9;33(3):459-64. doi: 10.1016/j.vaccine.2014.11.017. Epub 2014 Dec 8. PMID 25499651
- [Background] Thomas RE, Lorenzetti DL. Interventions to increase influenza vaccination rates of those 60 years and older in the community. Cochrane Database Syst Rev. 2018 May 30;5(5):CD005188. doi: 10.1002/14651858.CD005188.pub4. PMID 29845606